CLINICAL TRIAL: NCT04371315
Title: Risk Factors, Clinical Characteristics and Outcomes of Acute Infection With Coronavirus 2019 (COVID-19) In Children
Status: Recruiting | Type: Observational
Sponsor: St. Jude Children's Research Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: COVID-19
Record Dates: First submitted 2020-04-24; First posted 2020-05-01 (Actual); Last update posted 2025-11-10 (Actual); Status verified 2025-11

CONDITIONS: Corona Virus Infection; Pediatric Cancer; Adult Children; Cancer
MeSH Terms: conditions — Coronavirus Infections; Neoplasms

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Positive COVID-19: Baseline and Day 28: Respiratory and Whole blood Samples Collected, Days 7 and 14: Respiratory Samples Collected
  Monthly follow-up until Covid-19 is negative: Respiratory and Whole Blood Samples Collected
- Negative COVID-19: Baseline and Day 28: Respiratory and Whole blood Samples Collected, Days 7 and 14: Respiratory Samples Collected

SUMMARY:
Patient are being asked to provide respiratory and blood samples for a clinical research study because the patients have a virus called the novel coronavirus, or SARS-CoV-2, that causes the disease known as Covid-19.

Investigators do not know a lot about this virus, including all the ways it travels from person to person. Investigators also do not know if a person will get sick or not from the virus after being in close contact with someone who has the virus. Because of this, investigators are performing research on the virus found in respiratory secretions to get more information on how investigators can best detect and treat this new virus in the future.

Primary Objective

* To determine the clinical characteristics and outcomes of Covid-19 in children.
* To characterize the clinical risk factors of Covid-19 in children..

Secondary Objectives

* To characterize the immunological risk factors and serologic response to SARS-CoV-2 infection in children.- To evaluate the duration of viral shedding in children.
* To evaluate the duration of SARS-CoV-2 viral shedding in children. Exploratory Objective

DETAILED DESCRIPTION:
Nasal swabs will be collected from positive patient participants on Day 0. Timing of follow-up swabs will be guided by standard of care procedures.

Whole blood will be collected at Days 0. Follow-up blood sampling will be guided by standard of care procedures. Samples will be stored at -80oC.

Nasal swabs and whole blood will only be obtained at the same time standard of care procedures are performed. If a patient is not getting a blood draw, no sample will be collected.

ELIGIBILITY:
Patient Participant Inclusion Criteria:

* Less than 24 years old at the time of enrollment on study.
* St. Jude patients with laboratory confirmed Covid-19.

Exclusion Criteria:

* NA

Max Age: 24 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: All participants who meet eligibility criteria and consent to enrollment on the study.
Sampling Method: Non-Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2020-04-27 (Actual); Primary Completion 2025-12-01 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Characteristics and outcomes of acute respiratory infections due to COVID-19 in children. | Baseline-Day 60
  Clinical characteristics, including demographics, underlying diagnosis, and signs/symptoms, and outcomes, such as hospitalization, oxygen requirements, and mortality, will be summarized with counts and percentages.
Clinical risk factors of acute respiratory infection due to COVID-19 in children. | Baseline-day 60
  Pearson or Spearman's correlation of clinical risk factors such as age, underlying diagnosis, immunosuppression with outcomes as detailed in primary objective 1 will be evaluated.

SECONDARY OUTCOMES:
Immunologic response to acute respiratory infection due to COVID-19 in children. | Baseline-day 60
  Immunological (Absolute lymphocyte/monocyte counts (mm3) response measures, will be summarized with mean, standard deviation, median and range.
Immunologic response to acute respiratory infection due to COVID-19 in children. | Baseline-Day 60
  Immunological (Immunoglobulin level (mg/dL)) response measures, will be summarized with mean, standard deviation, median and range
Duration of viral shedding and evolution in children longitudinally. | Baseline-Day 60
  The duration of viral shedding, defined as the time between the first positive test date and the first negative test date, will be summarized for all participants with mean, standard deviation, median and range.

CONTACTS AND LOCATIONS:
Overall Officials: Diego Hijano, MD, Principal Investigator — St. Jude Children's Research Hospital
Locations (1):
- St. Jude Children's Research Hospital, Memphis, Tennessee, United States

REFERENCES:
- See also: St. Jude Children's Research Hospital — http://www.stjude.org
- See also: Clinical Trials Open at St.Jude — http://www.stjude.org/protocols